CLINICAL TRIAL: NCT03396107
Title: Role of Antenatal Corticosteroid Use in Elective Term Cesarean Section
Brief Title: Antenatal Corticosteroid in Elective Cesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Mostafa Haroun, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ACESC
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 6mg, IM, 48 hours before cesarean section
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo 6mg, IM, 48 hours before cesarean section
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 6mg, IM, 48 hours before cesarean section
  Arms: Dexamethasone
Drug: Placebo — Placebo 6mg, IM, 48 hours before cesarean section
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Caesarean section is a risk factor for the development of neonatal respiratory complications, mostly respiratory distress syndrome (RDS) and transient tachypnoea of the new-born, both in term and preterm infants.

DETAILED DESCRIPTION:
Infants born at term by caesarean delivery are more likely to develop respiratory morbidity than infants born vaginally, and this risk increases furthermore for the subgroup of children born by elective caesarean section, i.e. before onset of labour, with potentially severe implications. The risk is decreasing with advancing gestational age, and infants born between 37+0 and 37+6 weeks are at 1.7 times more risk for respiratory complications than those born between 38+0 and 38+6 weeks, which in turn are at 2.4 times more risk than the infants born between 39+0 and 39+6 weeks. If women were given two intramuscular injections of 12 mg of dexamethasone, two doses for 48 hrs,the rates of admissions were 5.2% at 37 weeks, 2.8% at 38 weeks, and 0.6% at 39 weeks. Although none of the babies in the control group died, admission will increase parental anxiety, the cost to nursery unit and invasive procedures including artificial ventilation giving mothers dexamethasone, two doses before elective section halved neonatal morbidity. Five studies lasting between three and 20 years with more than 1500 patients have shown no adverse effect of single course of antenatal corticosteroid, neither through infection of the fetus or mother nor in long term neurological or cognitive effect In view of this evidence, it is currently recommended that elective caesarean section should be deferred to 39 weeks. However approximately 10%-15% of woman planed for c/s may deliver before 38 weeks, and there may be concern on waiting in the presence of speci c indications or previous history. Respiratory morbidity in cases of term elective caesarean birth appears to have a different pathophysiology than in preterm birth, and retention in the lungs being the most likely cause.

Interestingly, recent evidence indicates that apart from the traditional mechanical concept of vaginal squeeze, molecular mechanisms (predominantly lung epithelial sodium channels promote alveolar uid drainage, and these channels are under active in fetuses unexposed to the process of labor. Glucocorticoid appears to increase the number and the function of thyroid hormones, providing a rational for their exogenous administration in cases of elective caesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age (18-35 years)
* Singleton pregnancy
* Gestational age (38-40 years)

Exclusion Criteria:

* Major maternal morbidities as DM and pre-eclampsia
* Sever oligohydramnios
* Premature rupture of membranes
* Women who receive steroids during pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 498 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory complications after cesarean section | 30 min
  To determine respiratory distress in infants born by elective cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fayek, Professor, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barber EL, Lundsberg LS, Belanger K, Pettker CM, Funai EF, Illuzzi JL. Indications contributing to the increasing cesarean delivery rate. Obstet Gynecol. 2011 Jul;118(1):29-38. doi: 10.1097/AOG.0b013e31821e5f65. PMID 21646928